CLINICAL TRIAL: NCT04211012
Title: A Phase II Study to Evaluate the Efficacy and Safety of Toripalimab Plus Nab-Paclitaxel With or Without Cisplatin as First-line Treatment of Unresectable Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: A Study on Toripalimab Plus Nab-Paclitaxel With or Without Cisplatin as First-line Treatment of Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Guo (Other)
Responsible Party: Sponsor-Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-UC-1015
Record Dates: First submitted 2019-11-22; First posted 2019-12-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — toripalimab

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Toripalimab plus Nab-Paclitaxel +/- cisplatin

INTERVENTIONS:
Drug: Toripalimab plus Nab-Paclitaxel +/- cisplatin — Toripalimab injection (JS001): 240mg, i.v.gtt, q3w; Nab-Paclitaxel: 260mg/m2, i.v.gtt, q3w Cisplatin: total dosage of 70 mg/m2 i.v.gtt, q3w，, complete all doses within the first 2 days of each cycle.
  Study treatment will be continued until disease progression or intolerable toxicity, or withdrawal at the discretion of the investigator or the subject, loss to follow-up, or initiation of other anti-cancer therapy, or death, whichever occurs first. Toripalimab will be administered no more than 2 years,and nab-paclitaxel with or without cisplatin will be administered up to 6 cycles.. If the subject is intolerable to cisplatin treatment according to the investigator's judgment, JS001 + Nab-Paclitaxel may be dosed.
  Dosing sequence: Toripalimab, Nab-Paclitaxel, cisplatin

SUMMARY:
This is a single-center, open-label，phase II study designed to evaluate the efficacy and safety of Toripalimab plus nab-paclitaxel with or without cisplatin as first-line treatment of unresectable locally advanced or metastatic urothelial carcinoma.Each enrolled Patient will receive Toripalimab plus nab-paclitaxel with or without cisplatin until progressive disease or intolerable toxicity occurs, then enter a survival follow-up period. Nab-paclitaxel with or without cisplatin will be administered for up to 6 cycles, and Toripalimab up to 2 years.

DETAILED DESCRIPTION:
Unresectable locally advanced or metastatic urothelial carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and are willing to sign informed consent form (ICF);
2. Age of ≥ 18 years at screening, male or female;
3. Histopathologically confirmed locally advanced (T4b, any N; or any T, N2-3) or metastatic (M1, stage IV) unresectable bladder urothelial carcinoma (including renal pelvis, ureter, bladder, urinary tract);
4. Not previously treated with systemic chemotherapy; Patients with urothelial carcinoma who have received prior adjuvant or neoadjuvant treatment or radiochemotherapy are eligible, provided that progression has occurred >6 months from last therapy (for radiochemotherapy and adjuvant treatment) or >6 months from last surgery (for neoadjuvant treatment).
5. At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
6. Providing tissue specimen for PD-L1 testing and related pathological report prior to enrollment for biomarker evaluation (tumor tissue specimen must be freshly obtained or archived within 3 months prior to enrollment; the fresh tissue must be a biopsy specimen of hollow needle punctured, excisedor resected);
7. ECOG performance status score of 0 or 1;
8. Life expectancy ≥ 12 weeks in the Investigator's opinion;
9. Adequate organ function:

   Hematology: absolute neutrophil count (ANC) ≥1.5×109/L; platelet count ≥100×109/L; hemoglobin ≥90g/L Renal: serum creatinine level ≤1.5 × ULN; urine protein ≤ 1+, if urine protein > 1 +, collect 24-hour urine protein determination, and the total amount should be ≤ 1 g,Liver: total bilirubin ≤ 1.5 × ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN; for patients with liver metastases, ALT and AST ≤ 5 × ULN Endocrine system: thyroid stimulating hormone (TSH) within normal range. Note: if the TSH is not within normal range at baseline, and T3 and free T4 are within normal range, the subject can still meet the inclusion criteria.

   Coagulation function: international normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless the subject is receiving anticoagulation therapy, PT or aPTT just needs to be within the expected therapeutic range of the anticoagulant).
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
11. Men of reproduction ability or women of pregnant possibility [amputation of uterus, bilateral oophorectomy or bilateral tubal ligation not performed, or prior to menopause (total menopause ≥1 year)] must adopt highly-effective contraceptive methods (e.g. oral contraceptives, intrauterine contraceptive device, abstinence of sexual intercourse or barrier contraception in combination with spermatocide) during the whole study, and continue contraception for 12 months after the last dose of study drug.

Exclusion Criteria:

1. Prior exposure to immune-mediated therapy (with the exclusion of Bacillus Calmette Guerin, BCG), including but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies, including therapeutic anticancer vaccines;
2. Currently participating in or having participated in another clinical study within 4 weeks prior to enrollment, unless it is an observational (non-interventional) clinical study;
3. Radiotherapy affect more than 30% of the bone marrow or extensive radiotherapy within 4 weeks prior to enrollment;
4. Major surgery within 4 weeks prior to enrollment;
5. Use of any live vaccines within 4 weeks before enrollment. Including but not limited to the following:mumps, rubella, measles, varicella/ herpes zoster (chicken pox), yellow fever, Rabies, Bacille Calmette-Guérin (BCG) and typhoid vaccine (inactivated virus vaccine allowed);
6. Treatment with immunosuppressive medications within 14 days prior to enrollment. The following are exceptions to this criterion:

   Intranasal, intraocular local steroids, or local steroid injections (eg, intraarticular injection) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Steroids as preventive medication for hypersensitivity reactions (eg, CT scan premedication)
7. Use of antineoplastic chemotherapy, biotherapy, hormone therapy or traditional herbal medicine t within 4 weeks prior to enrollment, except for the following:

   Concomitant medication of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable; Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable (eg, local radiotherapy or surgery);
8. History of (non-infectious) pneumonia/interstitial lung disease requiring steroid treatment, or ongoing pneumonia/interstitial lung disease requiring steroid treatment;
9. Uncontrolled concomitant diseases including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, arrhythmia, interstitial lung disease, or mental illness/social conditions consistent with the following characteristics: restricting study-specified compliance, significantly increasing the risk of developing AEs, or affecting patients' ability to provide informed consent form.
10. Known human immunodeficiency virus (HIV) infection (positive HIV antibody);
11. Active HBV or HCV infection; HBV DNA must be detected for patients with positive HbsAg or HBcAb at the screening; if HBV DNA test is positive at the same time (limit of quantitation 500 IU/ml, or reaching the positive value detected at the study center); Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
12. Active tuberculosis;
13. Allergies and adverse drug allergy reaction; Known hypersensitivity reactions to Toripalimab or any ingredient of Toripalimab Injection; History of serious hypersensitivity to nab-paclitaxel, cisplatin, or its preventive medication;
14. Subjects with active central nervous system (CNS) metastasis will be excluded. Patients who have prior therapies for brain or meningeal metastasis and has been stabilized for ≥ 3 months and has discontinued systemic steroids therapy (>10 mg/day prednisone or equivalent) > 4 weeks prior to enrollment could be included. If the CNS metastasis can be adequately treated and meet the requirement specified in the enrollment criteria, and the neurological symptoms can be recovered to ≤CTCAE grade 1 prior to enrollment (except the residual sign or symptom related with CNS treatment) for at least two weeks, the subject can participate in the study;
15. Active or previously recorded autoimmune or inflammatory diseases (including inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, etc.) within 2 years prior to enrollment. The following are exceptions to this criterion:

    Patients with vitiligo or alopecia; Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone (eg, treated Hashimoto's syndrome) or patients with psoriasis requiring no systemic treatment;
16. Having other malignant tumors that have not been recovered within past 5 years prior to enrollment, with the exception of those have been markedly cured, or curable cancer, such as skin basal cell carcinoma or squamous cell carcinoma, thyroid papillary carcinoma, localized low-risk prostate cancer, carcinoma in situ of cervix or breast; note: patients with localized low-risk prostate cancer (defined as ≤T2a stage, Gleason score ≤6 and PSA<10ng/mL at the diagnosis of prostate cancer (if measured) who have received radical therapy and have no biochemical recurrence of prostate specific antigen (PSA) can participate in this study);
17. Pregnant or lactating women;
18. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
19. History of any disease, therapy or abnormal laboratory examination that may confuse the study results, interfere with subject's participation in the whole study or not meet the best interest of subject's participation in the study, as judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | Up to 2 years
  ORR based on RECIST 1.1

SECONDARY OUTCOMES:
To evaluate Progression-free Survival (PFS) assessed by the investigator based on RECIST 1.1 criteria. | Up to 2 years
To evaluate Duration of Response (DOR) assessed by the investigator based on RECIST 1.1 criteria. | Up to 2 years
To evaluate Time to Response (TTR) assessed by the investigator based on RECIST 1.1 criteria. | Up to 2 years
To evaluate Disease Control Rate (DCR) assessed by the investigator based on RECIST 1.1 criteria. | Up to 2 years
To evaluate Overall Survival (OS) assessed by the investigator based on RECIST 1.1 criteria. | Up to 2 years
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment. | Up to 2 years
To evaluate the correlation between biomarkers (i.e. PD-L1, etc) and clinical endpoint (ORR) and/or incidence of adverse event. | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, No.52 Fucheng Road, Haidian District, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided